CLINICAL TRIAL: NCT03910881
Title: Technology-enabled Patient Support System for Self-management of Pediatric Cystic Fibrosis
Brief Title: Technology-enabled Patient Support System for Self-management of CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gabriela R Oates, Assistant Professor, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 300001749
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Perceived Stress Scale; Amyloid

STUDY DESIGN:
Intervention Model Description: Using a one-group pre-post design, evaluate the effect of the adapted technology-assisted PSS on patient-reported outcomes (PROs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open-platform patient support system (Experimental): Proof of concept testing of app
  Interventions: Other: Open-platform patient support system (PSS) app

INTERVENTIONS:
Other: Open-platform patient support system (PSS) app — The PSS app enables tracking and visualization of patient-selected health outcomes and sharing of select outcomes with family and providers. The CF clinical team and the family jointly decide which aspects of daily life to track, how often, and the content and frequency of patient-generated reports. Examples of daily care that can be tracked include symptoms (respiratory, gastrointestinal, pain), energy level, appetite, sleep, exercise, mood, medications, therapies, school/work attendance. Prior to a clinic visit, the patient/family generates a report of the outcomes they have been tracking, to help prepare for the visit and identify successes and areas of struggle. This information facilitates meaningful conversations during the visit and promotes shared decision-making. Patients/families can view their progress at any time and share selected outcomes with family and friends as often as desired.

SUMMARY:
This project will test a technology-enabled patient support system (PSS) as a self-management tool for children with CF and their family caregivers.

DETAILED DESCRIPTION:
The goal of this study is to refine and test a technology-enabled patient support system (PSS) as a tool for self-management of pediatric CF. The PSS includes two components: 1) patient-facing: an app with customizable dashboards for tracking patient-generated outcome measures and providing personally relevant decision-making support; and 2) clinic-based: clinical patient management and technical support. Using a one-group pretest-posttest design, we will evaluate the effect of the adapted technology-assisted PSS on patient-reported outcomes (PROs). Study hypothesis: Among pediatric CF patients treated at the UAB CF Center, the use of technology-aided PSS over 6 months will improve health-related quality of life (primary outcome) as well as patient satisfaction, patient activation, and shared decision-making (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Cystic Fibrosis -

Exclusion Criteria:

None

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (CFQ-R scores) | 3 months
  The primary outcome is difference in CFQ-R scores between pre/post intervention. The CFQ-R consists of 9 QOL domains (physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions) and 3 symptom scales (weight, respiratory, and digestion). Items for each CFQ-R domain are summed to generate a domain score ranging from 0 to 100, with higher scores indicating better QOL.
Health-related quality of life (CFQ-R scores) | 6 months
  The primary outcome is difference in CFQ-R scores between pre/post intervention. The CFQ-R consists of 9 QOL domains (physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions) and 3 symptom scales (weight, respiratory, and digestion). Items for each CFQ-R domain are summed to generate a domain score ranging from 0 to 100, with higher scores indicating better QOL.

SECONDARY OUTCOMES:
Shared decision-making (CollaboRate scores) | 3 months
  Difference in CollaboRate scores between pre/post intervention. CollaboRate includes 3 questions, each on a scale from 0-9, with higher scores indicating more shared decision-making.
Shared decision-making (CollaboRate scores) | 6 months
  Difference in CollaboRate scores between pre/post intervention. CollaboRate includes 3 questions, each on a scale from 0-9, with higher scores indicating more shared decision-making.
Patient/caregiver satisfaction (PACIC scores) | 3 months
  Difference in Patients' Assessment of Care for Chronic Conditions (PACIC) scores between pre/post intervention. PACIC includes 20 questions, each rated on a 5-point scale, with higher scores indicating higher quality of care.
Patient/caregiver satisfaction (PACIC scores) | 6 months
  Difference in Patients' Assessment of Care for Chronic Conditions (PACIC) scores between pre/post intervention. PACIC includes 20 questions, each rated on a 5-point scale, with higher scores indicating higher quality of care.
Patient/caregiver activation (PAM scores) | 3 months
  Difference in Patient Activation Measure (PAM) scores between pre/post intervention. PAM includes 13 questions, each with 4 response options, summed on a 0-100 scale, with higher scores indicating higher activation level.
Patient/caregiver activation (PAM scores) | 6 months
  Difference in Patient Activation Measure (PAM) scores between pre/post intervention. PAM includes 13 questions, each with 4 response options, summed on a 0-100 scale, with higher scores indicating higher activation level.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No